CLINICAL TRIAL: NCT06498297
Title: Analysis of the Impact of a Temporo-spatial Reorientation Tool on the Speed of Improvement of Confusional Syndrome, Assessed by the 4 "A" Test, in Patients Aged Over 75 Years Hospitalized in the Medical and Health Care Department. Geriatric Rehabilitation.
Brief Title: Analysis of the Impact of a Temporo-spatial Reorientation Tool on the Speed of Improvement of Confusional Syndrome
Acronym: Rob'Gazette
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9065
Record Dates: First submitted 2024-07-04; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Attention Disorder
Keywords: Attention Disorder; Confusion syndrome; Attentional disorders; Disorganization of cognitive functions
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Confusion syndrome is defined by attentional disorders and disorganization of cognitive functions that are acute and reversible. There are patient-specific predisposing factors and precipitating factors. Elderly people, due to their comorbidities, are more at risk. Confusion syndrome affects approximately 23% of elderly patients in the medical department, 33% in the rehabilitation department and its occurrence is preventable in 30 to 40% of cases. The health expenditure generated by its occurrence was estimated at 182 billion dollars per year by combining the expenditure of 18 European countries in 2011. The occurrence of a delirium increases the duration of hospitalization, increases the risk of falls, loss of autonomy, can lead to an impairment of quality of life at 6 months and is linked to excess mortality.

The gold standard for making the diagnosis of delirium is the use of the DSM-5 criteria, but their use is time-consuming and requires that staff be trained in their use. The 4 "A" test (tool to help identify confusional syndrome) can be used to monitor confusional syndromes; it has the advantage of being able to be taken in less than 3 minutes.

Concerning the management of a confusional syndrome, a non-pharmacological multi-component approach is recommended as first line for its prevention but there is no treatment to date. A tool to help with temporo-spatial reorientation (La Rob'Gazette) has been set up in the Medical Care and Geriatric Rehabilitation (SMRG) departments of the HUS

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 75 and over
* Hospitalized at the HUS in the SMRG department during the period from January 1, 2021 to April 31, 2023
* Passed at least a 4AT during hospitalization
* Absence of written opposition in the patient's medical file (and/or their legal representative if applicable) to the reuse of their data for scientific research purposes.

Exclusion Criteria:

- Presence of written opposition from the patient (and/or their legal representative if applicable) in their medical file.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patient aged 75 and over hospitalized at the HUS in the SMRG department during the period from January 1, 2021 to April 31, 2023 and havin passed at least a 4AT during hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04-24 (Estimated)

PRIMARY OUTCOMES:
Speed of improvement of the 4AT of the entire population | Up to 2 years
  The analysis will be undertaken on patients for whom at least two 4AT measurements are available (in order to be able to calculate a change). It will be based on a mixed linear model including the variable to be tested, time and their interaction. Variables deemed clinically relevant or statistically significant at the threshold of p < 0.10 will be included in a multivariate model. Then the non-significant and irrelevant variables will be removed from the model. The significance threshold will be 0.05 for this final model.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Soins de Soins Médicaux et de Réadaptation - CHU de Strasbourg - France, Strasbourg, France